CLINICAL TRIAL: NCT03976102
Title: A Double-blind, Parallel-group, Phase III Study to Compare the Efficacy, Safety, and Immunogenicity of Proposed Rituximab Biosimilar (DRL_RI) With MabThera® in Subjects With Previously Untreated (CD)20-Positive LTB Follicular Lymphoma
Brief Title: Compare Efficacy, Safety, and Immunogenicity of Proposed Rituximab Biosimilar (DRL_RI) With MabThera® in LTB Follicular Lymphoma
Acronym: FLINTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RI-01-006
Record Dates: First submitted 2019-04-15; First posted 2019-06-05 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; Dr. Reddy's Rituximab; Biosimilar (DRL_RI); FLINTER
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Clinical Phase III, randomised, multicentre, double-blind study to demonstrate the equivalence of DRL_RI to MabThera® in subjects with previously untreated, LTB-FL.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: DRL_RI (Experimental): DRL_RI (rituximab-Dr. Reddy's Lab) for infusion 375 mg/m2 administered via IV infusion on Days 1, 8, 15, 22 and Weeks 12, 20, 28 and 36
  Interventions: Biological: DRL_RI (Proposed rituximab biosimilar)
- Arm B: MabThera® (Active Comparator): MabThera® for infusion 375 mg/m2 administered via IV infusion on Days 1, 8, 15, 22 and Week 12, 20, 28 and 36.
  Interventions: Other: MabThera®

INTERVENTIONS:
Biological: DRL_RI (Proposed rituximab biosimilar) — Proposed rituximab biosimilar, 100mg and 500mg, concentrate for solution for infusion
  Arms: Arm A: DRL_RI
Other: MabThera® — Reference product rituximab, 100mg and 500mg, concentrate for solution for infusion
  Arms: Arm B: MabThera®

SUMMARY:
The primary objective of the current study is to demonstrate the equivalent efficacy of rituximab (DRL_RI) and MabThera® in subjects with Low Tumor Burden Follicular Lymphoma (LTB-FL).

Also evaluated by Pharmacokinetic, safety, and immunogenicity assessment between a proposed biosimilar (DRL_RI) and the RMP, as an component of clinical study program, and collectively providing the evidence of biosimilarity.

The study will compare the safety and efficacy of DRL_RI vs MabThera in patients with Low Tumor Burden Follicular Lymphoma (LTB-FL). The primary objective is to establish comparative efficacy as measured by ORR up to week 28

DETAILED DESCRIPTION:
It is planned to randomise approx. 312 subjects at approximately ≥ 130 study sites worldwide. Subjects with LTB-FL will be randomized to receive either DRL_RI or MabThera®. Till date, 68 patients have been randomized for the study.

The study specific objectives are mentioned below:

Primary Objective:

• To demonstrate the equivalent efficacy of DRL_RI (biosimilar rituximab) and MabThera in subjects with CD20-positive, LTB FL, as measured by overall response rate (ORR) up to Week 28 evaluated in accordance with Cheson, 1999 response criteria for Non-Hodgkin's Lymphomas.

Secondary Objectives:

* To compare the progression-free survival (PFS), overall survival (OS), and duration of response (DOR) of DRL_RI with MabThera® in subjects with CD20-positive, LTB FL.
* To compare the safety, tolerability, and immunogenicity of DRL_RI with MabThera in subjects with CD20-positive, LTB-FL.

Exploratory Objectives

* To explore the pharmacokinetic (PK) parameters of DRL_RI and MabThera, using a population-PK modelling approach.
* To explore the pharmacodynamic parameters of DRL_RI and MabThera.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is Male or female subjects aged ≥18 years of age.
2. Subject is histologically confirmed, Grade 1-3a, previous ly untreated, CD20-pos itive.
3. Subject has Ann Arbor Stage II to IV and ECOG status of 0 to 1.
4. Subject has Low tumor burden follicular lymphoma as per Groupe d'Etude des Lymphomes Folliculaires (GELF) Criteria
5. Subject has at least 1 measurable tumor mass in 2 dimensions, and the mass must be:

   1. Nodal lesion >15 mm in the longest dimension; or
   2. Noda l lesion >10 mm to he longest dimension; dimens ion and >10 mm in the shortest dimension; or
   3. Extra-nodal lesion with both long and short dimensions ≥10 mm.
6. Subject has Life expectancy ≥3 months.
7. If female subject, then subject should be non-pregnant, non-lactating.

Exclusion Criteria:

1. Subject with prior use of rituximab or any CD20 monoclonal antibody for any reason.
2. Subjects with known hypersensitivity to rituximab or its excipients, or to proteins of murine or other foreign origin.
3. Any prior therapy for follicular lymphoma (including but not limited to chemotherapy, radiotherapy) or subjects on chronic supra-substitutive doses of systemic gluco-corticosteriods.
4. Subjects who, in the opinion of the Investigator, require additional concomitant treatment for lymphoma.
5. Evidence of histologic transformation to high grade lymphoma or diffuse large B-cell lymphoma.
6. Subjects with known sero-positivity for or history of active viral infection with human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) will be excluded. And if positive for hepatitis B core antibody or hepatitis C virus (HCV) antibody can only be enrolled if HBV - DNA level <20 IU/mL (or 112 copies/mL) and HCV - RNA is negative respectively by PCR test..
7. Subjects who have received a live vaccine within last 3 months of the first administration of study drug.
8. Subjects with history or presence of a medical condition or disease that in the Investigator's opinion would place the subject at an unacceptable risk for study participation.
9. Participation in any clinical study or having taken any investigational therapy (within 2-months of the first dose of study drug.
10. Women of childbearing potential who do not consent to use highly effective methods of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliso Sopia, MD, Study Director — Parexel
Locations (4):
- United States (4):
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - University of Tennessee Medical Center - Cancer Institute, Knoxville, Tennessee
  - Gulf coast Oncology Associates, PA, Houston, Texas

REFERENCES:
- [Derived] Maharaj N, Uppada DR, Eswaraiah A, Kakkattu R, Reddy P, Kalenik VA, Belada D, Ramos AO, Kim JS, Baranau YV. Efficacy and safety of rituximab biosimilar (DRL_RI) versus MabThera(R) in low-tumor-burden follicular lymphoma: the FLINTER study. Ther Adv Med Oncol. 2025 May 24;17:17588359251339925. doi: 10.1177/17588359251339925. eCollection 2025. PMID 40421128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 4 sites in the United States from 15 May 2019 to 27 February 2023. The final participant was examined or received an intervention for the purposes of final collection of data for the primary outcome on 28 September 2022.
Pre-assignment Details: All the assessments were performed as per the schedule of the assessments.
Groups:
- Arm A: DRL_RI: Randomized participants were administered rituximab biosimilar-Dr. Reddy's Lab (DRL_RI) 375mg/m^2 via intravenous (IV) infusion on Days 1, 8, 15, 22 and Weeks 12, 20, 28 and 36.
- Arm B: MabThera®: Randomized participants were administered MabThera® 375 mg/m^2 via IV infusion on Days 1, 8, 15, 22 and Weeks 12, 20, 28 and 36
Period: Overall Study
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Started | 162 | 155
Completed | 143 | 129
Not Completed | 19 | 26
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Adverse Event | 2 | 4
Not completed — Not related to Covid-19 | 9 | 13
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 3 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Analysis Set included all randomized participants.
Groups:
- Arm A: DRL_RI: Randomized participants were administered DRL_RI 375 mg/m^2 via IV infusion on Days 1, 8, 15, 22 and Weeks 12, 20, 28 and 36
- Total: Total of all reporting groups
Arm/Group | Arm A: DRL_RI | Arm B: MabThera® | Total
Number analyzed (Participants) | 162 | 155 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (12.37) | 55.8 (13.03) | 56.7 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 78 | 160
  Male | 80 | 77 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 118 | 110 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 104 | 107 | 211
  Asian | 51 | 46 | 97
  Black or African American | 0 | 0 | 0
  Aboriginal/Torres Strait Islander | 1 | 0 | 1
  Unknown | 1 | 1 | 2
  Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR) for Low Tumor Burden Follicular Lymphoma
Description: Best Overall Response Rate (BORR) is defined as the proportion of participants in each treatment group that achieved a best overall response of either Complete response (CR), unconfirmed Complete response (CRu) or Partial response (PR), up to Month 7 (Week 28) based on central radiology review in accordance with the Cheson, 1999 response criteria for Non-Hodgkin's Lymphomas. As per Cheson 1999, response criteria for target lesions and assessed by radiology: Complete response (CR): All lesions with a longest diameter should be regressed to normal size (≤ 15 mm) or short axis regressed to ≤ 10 mm with confirmed Bone marrow normalization; unconfirmed Complete response (CRu): All lesions with a longest diameter should be regressed to normal size (≤ 15 mm) or short axis regressed to ≤ 10 mm with non-confirmed Bone marrow normalization; Partial Response (PR): ≥ 50 % decrease of sum of products of diameter(SPD) of all the target lesions; Overall Response (OR)=CR+CRu+PR.
Time Frame: Month 7 (Week 28)
Population: The ITT Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm A: DRL_RI: Randomized participants were administered DRL_RI 375mg/m^2 via IV infusion on Days 1, 8, 15, 22 and Weeks 12, 20, 28 and 36.
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 155
percentage of participants | 80.2 [73.3 to 86.1] | 79.4 [72.1 to 85.4]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) is defined as proportion of participants in each treatment group achieved a complete response or partial response at week 12 and week 28 based on central radiology review in accordance with published response criteria for malignant lymphoma. As per Cheson 1999, response criteria for target lesions and assessed by radiology: Complete response (CR): All lesions with a longest diameter should be regressed to normal size (≤ 15 mm) or short axis regressed to ≤ 10 mm with confirmed Bone marrow normalization; unconfirmed Complete response (uCR): All lesions with a longest diameter should be regressed to normal size (≤ 15 mm) or short axis regressed to ≤ 10 mm with non-confirmed Bone marrow normalization; Partial Response (PR): ≥ 50 % decrease of sum of products of diameter(SPD) of all the target lesions; Overall Response (OR)=CR+uCR+PR.
Time Frame: Week 12, Week 28
Population: The ITT Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 155
percentage of particpants
  Week 12 | 62.3 [54.4 to 69.8] | 63.9 [55.8 to 71.4]
  Week 28 | 75.3 [67.9 to 81.7] | 73.5 [65.9 to 80.3]

3. Secondary Outcome: Complete Response Rate
Description: Complete Response rate is defined as the proportion of participants in each treatment group who achieved complete response up to particular visit based on investigator assessment in accordance with the response criteria for malignant lymphoma. As per Cheson 1999, response criteria for target lesions and assessed by radiology: Complete response (CR): All lesions with a longest diameter should be regressed to normal size (≤ 15 mm) or short axis regressed to ≤ 10 mm with confirmed Bone marrow normalization.
Time Frame: Week 28
Population: The ITT Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 155
percentage of participants | 32.7 [25.6 to 40.5] | 34.2 [26.8 to 42.2]

4. Secondary Outcome: Complete Response Rate as a Best Response
Description: Complete Response Rate as a Best Response is defined as the proportion of participants in each treatment group that achieved the best complete response up to Week 28 based on central radiology review in accordance with the Cheson 1999, response criteria for malignant lymphoma. As per Cheson 1999, response criteria for target lesions and assessed by radiology: Complete response (CR): All lesions with a longest diameter should be regressed to normal size (≤ 15 mm) or short axis regressed to ≤ 10 mm with confirmed Bone marrow normalization.
Time Frame: Week 28
Population: The ITT Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 155
percentage of participants | 34.0 [26.7 to 41.8] | 35.5 [28.0 to 43.6]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) defined as the time from date of the first documentation of tumor response (Complete Response, unconfirmed complete response or partial response) to the date of first documentation of progressive disease (PD) or to death due to any cause up to 52 weeks/ End of study (EOS). Progression is defined as per Cheson 1999, response criteria is:
  Target Nodal SPD Progression: at least one node must be abnormal, and the SPD of all nodes must increase by ≥ 50% from its nadir SPD.
  Target Extranodal SPD Progression: at least one extranodal lesion must be present and the SPD of all extranodal lesions must increase by ≥ 50% from its nadir SPD.
  Also, if a patient had any unequivocal progression in non-target lesions; and detection of any new nodal lesion (longest diameter [LDi] 15mm with an absolute increase of 5mm) his/her response was considered as Progressive disease.
Time Frame: Week 52
Population: The ITT Analysis Set included all randomized participants. The number analyzed are the participants with complete response, unconfirmed complete response or partial response.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Arm A: DRL_RI: Randomized participants were administered DRL_RI 375mg/m^2 via intravenous (IV) infusion on Days 1, 8, 15, 22 and Weeks 12, 20, 28 and 36.
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 134 | 130
Weeks | NA [NA to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study. | NA [NA to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study.

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from date of randomization to the date of documented progressive disease or death due to any cause. Progression is defined as per Cheson 1999, response criteria is:
  Target Nodal SPD Progression: at least one node must be abnormal, and the SPD of all nodes must increase by ≥ 50% from its nadir SPD.
  Target Extranodal SPD Progression: at least one extranodal lesion must be present and the SPD of all extranodal lesions must increase by ≥ 50% from its nadir SPD.
  Also, if a patient had any unequivocal progression in non-target lesions; and detection of any new nodal lesion (LDi 15mm with an absolute increase of 5mm) his/her response was considered as Progressive disease.
Time Frame: Week 52
Population: The ITT Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 155
Weeks | NA [NA to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study. | NA [NA to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study.

7. Secondary Outcome: Overall Survival (OS)
Description: The Overall survival (OS) defined as the time from date of randomization to the date of death from any cause up to 52 weeks or EOS.
Time Frame: Week 52
Population: The ITT Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 155
Weeks | NA [NA to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study. | NA [NA to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study.

8. Secondary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of DRL_RI and MabThera® in participants with CD20-positive, LTB-FL was evaluated.
Time Frame: From Screening (Day -28 to -1) up to 52 weeks
Population: The Safety Analysis Set (SAF) will include all the participants who have received at least one dose of study drug. The SAF will be used for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 162 | 153
Participants
  Treatment-emergent adverse events (TEAEs) | 113 | 103
  Non-TEAEs | 13 | 18
  Infusion related AEs | 28 | 32
  TEAE>=Common terminology Criteria for Adverse events (CTCAE) grade 3 | 30 | 24
  Serious TEAEs | 22 | 21
  TEAEs related to study drug | 48 | 50
  Fatal TEAEs | 3 | 2

9. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA)
Description: The immunogenicity of the Proposed Rituximab Biosimilar (DRL_RI) with MabThera® among trial participants was compared.
Time Frame: On Day 1, Week 2, Week 3, Week 4, Week 12 post dose
Population: The ITT Analysis Set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
Number analyzed (Participants) | 48 | 41
Participants
  Day 1 | 2 | 0
  Week 2 | 2 | 0
  Week 3 | 1 | 0
  Week 4 | 2 | 0
  Week 12 | 2 | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -28 to -1) up to 52 weeks
Description: The SAF include all participants who have received at least 1 dose of study drug and will be used for safety analysis. The number of participants analyzed for safety analysis is different from ITT analysis population (ITT population was defined as all patients randomized). Two participants were randomized but did not receive the treatment with MabThera and therefore were not included in the SAF but included in ITT.
Arm/Group | Arm A: DRL_RI | Arm B: MabThera®
All-Cause Mortality (participants affected / at risk) | 3/162 | 2/153
Serious Adverse Events (participants affected / at risk) | 22/162 | 21/153
Other Adverse Events (participants affected / at risk) | 47/162 | 49/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: DRL_RI (N=162) | Arm B: MabThera® (N=153)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 10 (10) | 5 (5)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Infusion-related reaction (Investigations) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: DRL_RI (N=162) | Arm B: MabThera® (N=153)
Neutropenia (Blood and lymphatic system disorders) | 13 (14) | 2 (3)
Nausea (Gastrointestinal disorders) | 6 (8) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 8 (10)
Pyrexia (General disorders) | 1 (1) | 10 (10)
COVID-19 (Infections and infestations) | 19 (20) | 17 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (14) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03976102/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03976102/SAP_001.pdf